CLINICAL TRIAL: NCT00626314
Title: A Multi-Center, Double-Blind, Randomized, Placebo Controlled, Trial to Assess the Efficacy, Safety and Tolerability of Transplanting Autologous Skeletal Myoblasts, Into Infarcted Myocardium, Using an Endomyocardial Delivery System
Brief Title: Study to Assess the Efficacy and Safety of Transplanting Autologous Skeletal Myoblasts, Into Infarcted Heart, Using an Catheter Delivery System
Acronym: CAuSMIc II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mytogen, Inc. (Industry)
Responsible Party: JONATHAN DINSMORE, PHD/SENIOR VICE PRESIDENT, CLINICAL&REGULATORY AFFAIRS, MYTOGEN/ADVANCED CELL TECHNOLOGY
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDAM06-5
Record Dates: First submitted 2008-02-21; First posted 2008-02-29 (Estimated); Last update posted 2008-02-29 (Estimated); Status verified 2008-02

CONDITIONS: Ischemic Cardiomyopathy
MeSH Terms: interventions — salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (2):
- 1 (Experimental): myoblast
  Interventions: Biological: myoblast
- 2 (Sham Comparator): sham injection procedure
  Interventions: Biological: sham

INTERVENTIONS:
Biological: myoblast — autologous myoblast
  Arms: 1
Biological: sham — sham injection procedure
  Arms: 2

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of injecting myoblasts (grown from your own skeletal muscle), using a catheter device, directly into the damaged heart muscle for treatment of severe heart failure.

DETAILED DESCRIPTION:
Given the limited treatment options available to patients with congestive heart failure, there is a need for alternative therapies. Autologous skeletal myoblast transplantation has been demonstrated in pre-clinical studies to be a safe and effective treatment of heart failure. Initial clinical studies have shown that autologous myoblasts can be delivered into infracted myocardium by both direct epicardial and endomyocardial injection. However, autologous skeletal myoblast transplantation via percutaneous endomyocardial injection has the potential to play a significant role in such congestive heart failure patients without the need for surgical risk and general anesthesia. Thus, a Phase 2 clinical trial is proposed in order to evaluate the effectiveness of autologous myoblast delivered by endomyocardial injection for the treatment congestive heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects with ischemic cardiomyopathy and previous myocardial infarction
2. New York Heart Association Classification III - ambulatory Class IV
3. Ejection fraction < 35% as determined by any method at baseline evaluation
4. Subjects could be considered for enrollment if CRT placement has occurred greater than three months previously with no clinical improvement, CRT settings are judged to be optimized and the subject continues to meet all other inclusion criteria (inadequate-responders).
5. Documentation of ineligibility for coronary revascularization and/or valve repair/ replacement by review of recent left heart catheterization (within six months of baseline).
6. Receiving optimally tolerated doses of standard, stable pharmacotherapy, including angiotensin-converting enzyme inhibitors, unless intolerant or contra-indicated, diuretics, ß-receptor blockers for at least one month prior to enrollment
7. Severe myocardial perfusion abnormality documented by SPECT imaging, involving at least 1/3 of a vascular territory, as confirmed by core lab.

Exclusion Criteria:

1. Age < 21 years or > 75 years.
2. Significant coronary stenosis, as determined by the Investigator, which may potentially require percutaneous or surgical revascularization within 12 weeks of enrollment.
3. Recent (within 4 weeks), documented acute coronary syndrome, i.e. (Q wave or non-Q wave infarction) or hospitalization for unstable angina.
4. Documented cerebrovascular accident (stroke) or TIA within 60 days.
5. Left ventricular thrombus (mobile or mural-based) as evidenced by ventriculogram or echocardiography.
6. Clinically significant electrocardiographic abnormalities that may interfere with subject safety during the intracardiac mapping and injection procedure. Patients with right bundle branch block with basal septal infarction.
7. Subjects with CRT placement within three months of enrollment or intent to insert CRT, or CRT settings not judged to be optimized
8. High grade atrioventricular block not corrected by permanent pacemaker or ICD.
9. Frequent or recurrent, ventricular tachycardia in absence of an ICD.
10. Atrial fibrillation with uncontrolled ventricular response
11. Significant uncorrected valvular disease, which results in additional hemodynamic compromise and/or would require valvular repair or replacement. Patients with severe aortic stenosis or status-post mitral or aortic mechanical valve replacement.
12. Severe peripheral vascular disease, such that femoral access would be prohibited.
13. INR > 1.5 in absence of coumadin or partial thromboplastin time (PTT) >20% above ULN, or thrombocytopenia (platelet count < 75,000).
14. Significant renal dysfunction (e.g., creatinine >2.5 mg/dL) or liver disease (e.g., serum glutamic-oxaloacetic transaminases / aspartate aminotransferase SGOT/AST or serum glutamic-pyruvic transaminases/alanine aminotransferase SGPT/ALT > 4 x upper limit of normal [ULN]).
15. Currently enrolled, or have been enrolled within 30 days, in another investigational drug or device study that has not completed the protocol required follow-up period.
16. Subjects who have received a prior investigational stem cell or angiogenic agent.
17. Subjects who have tested positive for Human Immunodeficiency Virus (HIV), Hepatitis B Virus (HBV), and/or Hepatitis C Virus (HCV).
18. History of skeletal muscle disease, e.g. family history of acute or chronic skeletal muscle disease including infectious, drug-induced, familial, autoimmune and idiopathic myopathies.
19. Creatine phosphokinase (CK) or lactate dehydrogenase elevated greater than three times normal or unexplained elevations of CK.
20. Female subjects who are pregnant or nursing or any subject with reproductive capabilities unwilling to use effective birth control for the duration of the study period.
21. Evidence of concurrent infection of any type (e.g. Elevated white blood cell count {WBC>13,000}, temperature of >38.5 C, or infiltrate on chest x-ray).
22. Any other major illness, which, in the Investigator's judgment, will interfere with the subject's ability to comply with the protocol, compromises subject safety, or interferes with the interpretation of the study results.
23. Idiopathic Cardiomyopathy, hypertrophic cardiomyopathy
24. Subjects with ventricular wall thickness in the infarct zone of < 5 mm measured by echocardiogram at baseline.
25. Patients on chronic (or chronic intermittent) IV inotropic medication. -

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Estimated)
Dates: Start 2008-03; Primary Completion 2010-03 (Estimated); Study Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Kansas City Cardiomyopathy Questionnaire | 6 months

SECONDARY OUTCOMES:
Cardiovascular mortality | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Mercy Gilbert, Gilbert, Arizona, United States